CLINICAL TRIAL: NCT06732661
Title: A Prospective Randomized Controlled Study on the Impact of Preserving the Pre-cardial Fat Pad During Sleeve Gastrectomy on Postoperative Gastroesophageal Reflux
Brief Title: Preserving the Pre-cardial Fat Pad During Sleeve Gastrectomy on Postoperative Gastroesophageal Reflux
Acronym: Pad and SG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fat pad-SG; 82070685 (Other Grant/Funding Number: National Natural Science Foundation of China (General Program))
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-07

CONDITIONS: Sleeve Gastrectomy; Pre-cardial Fat Pad; Excessive Weight Loss; Total Weight Loss; Gastroesophageal Reflux Disease
Keywords: sleeve gastrectomy; pre-cardial fat pad; Gastroesophageal Reflux Disease; Weight Loss
MeSH Terms: conditions — Gastroesophageal Reflux; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preserve pre-cardial fat pad (No Intervention): For this group, a sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. A security distance of 10 mm lateral to the esophagus is respected without dissection of pre-cardial fat pad.
- Dissect pre-cardial fat pad (Experimental): For this group, a sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. Dissect the pre-cardial fat pad, and a security distance of 10 mm lateral to the esophagus is respected.
  Interventions: Procedure: Preserve pre-cardial fat pad; Procedure: Dissect pre-cardial fat pad

INTERVENTIONS:
Procedure: Preserve pre-cardial fat pad — For this group, a sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. A security distance of 10 mm lateral to the esophagus is respected without dissection of pre-cardial fat pad.
  Arms: Dissect pre-cardial fat pad
Procedure: Dissect pre-cardial fat pad — For this group, a sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. Dissect the pre-cardial fat pad, and a security distance of 10 mm lateral to the esophagus is respected.
  Arms: Dissect pre-cardial fat pad

SUMMARY:
Gastroesophageal reflux disease (GERD) is one of the most common chronic conditions that can affect one's quality of life. Laparoscopic sleeve gastrectomy (LSG) has become a popular technique and currently is the most frequently practiced surgical operation to treat obesity today. However, the prevalence of GERD following SG can be fairly high. Several studies have noted an incidence between 6% and 47%.

The angle of His is important for the maintenance of esophageal anti-reflux ability, and prevent GERD. Most SG operating consensus recommends surgeons should stay at least 1 cm away from the angle of His. However, on consensus was reached about the pre-cardial fat pad should be routinely dissected or not to avoid leaving behind a large fundus consensus.

The investigators propose to perform a prospective randomized controlled study to dissect the pre-cardial fat pad or not in obese patients followig sleeve gastrectomy to prevent GERD.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is one of the most common chronic conditions that can affect one's quality of life. Laparoscopic sleeve gastrectomy (LSG) has become a popular technique and currently is the most frequently practiced surgical operation to treat obesity today. However, the prevalence of GERD following SG can be fairly high. Several studies have noted an incidence between 6% and 47%.

The angle of His is important for the maintenance of esophageal anti-reflux ability, and prevent GERD. Most SG operating consensus recommends surgeons should stay at least 1 cm away from the angle of His. However, on consensus was reached about the pre-cardial fat pad should be routinely dissected or not to avoid leaving behind a large fundus consensus.

The dissection of pre-cardial fat pad is helpful to fully expose the gastric fundus, to accurately judge the distance between the incision line and the esophagus, and to help the suture embedding of the incision line. However, the disadvantages might increase the rate of GERD. While retaining the pre-cardial fat pad may contribute to the reduction of GERD rate. However, it might not be conducive to the judgment of cutting distance to the esophagus and the procedure of suture embedding. Futhermore, there may be gastric fundus residue during SG.

The investigators propose to perform a prospective randomized controlled study to dissect the pre-cardial fat pad or not in obese patients followig sleeve gastrectomy to prevent GERD.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 32.5 kg/m2 with or without T2DM;
* 27.5 kg/ m2 < BMI < 32.5 kg/m2 with T2DM but failed conservative treatment and combined with at least two metabolic diseases or comorbidities;
* Duration of T2DM ≤15 years with fasting Cpeptide ≥ 50% of normal lower limit
* Waist circumference: male ≥ 90 cm, female ≥ 85 cm
* Age within 16~65 years old

Exclusion Criteria:

* GERD preoperatively
* Hiatus hernia approved by gastroscopy preoperatively
* Pregnancy;
* A history of mental illness and neurological disease;
* The patient refuses surgery;
* Combined with pituitary tumor;
* Long-term use of antidepressant drugs;
* Long-term use of immunosuppressants;
* Situations in which the investigator or other examiner considers from the enrolled study that there are good reasons for nonconformity: if there are potential inconsistencies with the clinical protocol

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of gastroesophageal reflux disease | 1 year
  The rate of gastroesophageal reflux disease following sleeve gastrectomy at 1 year

SECONDARY OUTCOMES:
Complications | 30 days postoperatively
  Complications within 30 days postoperatively
Operating time | During the operation
  Time from opeing of the operation to the end of the operation
excessive weight loss | 3 months, 6 months, 1 year postoperativel
  Percentage of excess weight loss (EWL) at any time postoperative was calculated as the amount of weight loss divided by the amount of excess weight times 100%.
total weight loss | 3 months, 6 months, 1 year postoperatively
  total weight loss compared with preoperative weight

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No